CLINICAL TRIAL: NCT02681276
Title: Clinical and Microbiological Evaluation of 0.5% Versus 3% Sodium Hypochlorite in Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Thomas Kvist, Clinical Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Irrigation 3% NaOCl
Record Dates: First submitted 2016-01-26; First posted 2016-02-12 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Pulpitis; Apical Periodontitis
Keywords: Irrigation during root canal treatment; Sodium Hypochlorite
MeSH Terms: conditions — Pulpitis; Periapical Periodontitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irrigation with 3% NaOCl (Experimental): After informed consent the patient was randomly assigned to have the root canal treatment performed with a 3 % NaOCl irrigation during instrumentation. If the patient's first visit was on an uneven date the concentration of the irrigant was 3 %.
  Interventions: Procedure: Irrigation with 3% NaOCl
- Irrigation with 0.5% NaOCl (Active Comparator): After informed consent the patient was randomly assigned to have the root canal treatment performed with a 0.5 % NaOCl irrigation during instrumentation. If the patient's first visit was on an even date the concentration of the irrigant was 0.5 %.
  Interventions: Procedure: Irrigation with 0.5% NaOCl

INTERVENTIONS:
Procedure: Irrigation with 3% NaOCl — All the operators are informed to perform the endodontic treatment the way they normally do. The only variation during treatment was the concentration of the sodium hypochlorite solution for irrigation of the root canal.
  Arms: Irrigation with 3% NaOCl
Procedure: Irrigation with 0.5% NaOCl — All the operators are informed to perform the endodontic treatment the way they normally do. The only variation during treatment was the concentration of the sodium hypochlorite solution for irrigation of the root canal.
  Arms: Irrigation with 0.5% NaOCl

SUMMARY:
Aim: To compare the clinical antimicrobial and adverse effects of irrigation with Sodium Hypochlorite (NaOCl) 0.5% versus NaOCl 3% during root canal treatment.

Methodology: Consecutive patients referred to a specialist clinic of endodontics are randomly assigned to have the root canal treatment performed with a concomitant irrigation either with a buffered 0.5 % NaOCl (Dakin's solution) or 3 % NaOCl. Teeth with vital or necrotic pulps and retreatment cases were included. Root canal treatment procedures varied but followed the routines of the Specialist Clinic of Endodontics, Public Dental Health, Gothenburg, Sweden. Immediately before the root canal filling a microbial sample is taken from the operative field and the root canal. The bacterial samples were processed at the laboratory as outlined by Möller (1966). After each visit each patient was instructed to fill in a questionnaire and assess his or her post-operative pain on a visual analogue scale (VAS), with endpoints 0= "no pain" and 10= "worst imaginable pain", for seven consecutive days. The Fischer's exact test was used for statistical analyses of the differences in outcome between the groups.

DETAILED DESCRIPTION:
The aim of the present study is to compare the antimicrobial and immediate clinical effect of NaOCl 0.5% with the effect of NaOCl 3% in the endodontic treatment of teeth referred to the Specialist Clinic of Endodontics, Göteborg, Public dental Health, Västra Götaland. The efficiency of the treatment will be evaluated with sampling and cultivation methods and the assessment of patients' symptoms with a visual analogue scale.

The sample size calculation was performed with a type I error of 0.05 and statistical power of 80 %. The investigators expected 70 % of the samples to be free from bacteria growth in the control group and the investigators considered clinically relevant a difference of 15 % between the groups in order to demonstrate significant differences attributable to the experimental therapy used. The investigators want our sample size to be two hundred sixty four patients, 132 to each group.

A detailed explanation of the purpose of the study was given. Patients were also informed about the confidentiality of the data to be collected and about the voluntary participation. Every patient gets assigned a code that indicates which group they belong so the same irrigant is used in case of more than one visit.

Root canal treatment followed the standard principles of the Specialist Clinic of Endodontics, Göteborg, Public dental Health, Västra Götaland but the treatments were not restricted to a single protocol.

The recommended minimum or optimal apical size of canal preparation is size 25. All the operators are informed to perform the endodontic treatment the way operators normally do. The only variation during treatment was the concentration of the sodium hypochlorite solution for irrigation of the root canal. One group was irrigated with Sodium Hypochlorite 0.5 % (Dakin's solution) and the other group with Sodium Hypochlorite 3 %.

Operators were free to choose any additional irrigant as clinically perceived necessary. The irrigants available at the clinic were 17% ethylene-diamine-tetra-acetic acid (EDTA) and iodine-potassium-iodide (IPI) 5% used as a short duration antimicrobial agent as intracanal medication for 10 minutes.

Canal irrigation was carried out using 27 gauge side-cut open end needles (Monoject Luer lock syringe) with supplementation by ultrasonic agitation. Calcium hydroxide was the standard inter-appointment medicament. After sampling procedures gutta-percha and AH-plus sealer were used for root filling.

The access cavity was filled with Intermediate Restorative Material (IRM) or a permanent filling with composite after each appointment and after finished root canal treatment.

After bacterial sampling of the root canal, the samples were processed at the laboratory as outlined by Möller. Anaerobic incubation was done in a semi liquid medium (Hunton medium) inoculated under flow of oxygen-free gas. The mediums are checked daily for 14 days or until there is signs of microbial growth.

Fischer's exact test will be used for comparisons between groups regarding growth / no growth. For assessments of pain on the VAS t-test and 95% confidence intervals will be used. All hypothesis tests will be conducted at the 0.05 level of significance.

The outcomes will be analysed in term of positive Cultures and post operative pain. This is discussed further elsewhere in this application.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of and willing to have a root canal treatment
* Diagnosis Pulpitis
* Diagnosis Apical periodontitis.
* If a patient was referred for more than one tooth just the first treated tooth was included in the study.
* The teeth had to be restorable and placement of rubber dam must be possible.

Exclusion Criteria:

* patient does not understand Swedish
* the tooth will be treated with a retrograde approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2014-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Assessing bacterial growth in the root canal (positive meaning cultivable bacteria present, negative meaning absence of cultivable bacteria) | Sample from the root canal taken immediately before root canal filling, assessing growth for 30 days after the sample is taken.
  Bacterial sampling was taken just before the root canal filling. The sodium hypochlorite solution and the iodine-potassium-iodide were inactivated with 5 % sodium thiosulfate solution for 30 sec. The canals were then filled with VMGA I, dentinal shavings were produced with H files ISO #25. The entire canal content was absorbed by means of charcoal points and transferred to VMGA III.

SECONDARY OUTCOMES:
Assessment of post-operative pain using a questionnaire containing 7 visual scales. | 7 consecutive days after each appointment
  Each patient was instructed to fill in a questionnaire after each visit. This questionnaire contains seven visual scales (VAS) based on a 10 cm line determining the pain level. The patient is asked to estimate the pain they have 7 days after the endodontic procedure where 1 is very mild pain and 10 the worse pain they can imagine. The questionnaires were measured with a plastic ruler and the recordings will be transposed to numbers and registered in the excel file by the main investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kvist, phD, Study Chair — Göteborg University
Locations (1):
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
The data is going to be published at a Group level

REFERENCES:
- [Background] Spencer HR, Ike V, Brennan PA. Review: the use of sodium hypochlorite in endodontics--potential complications and their management. Br Dent J. 2007 May 12;202(9):555-9. doi: 10.1038/bdj.2007.374. PMID 17496870
- [Result] Ayhan H, Sultan N, Cirak M, Ruhi MZ, Bodur H. Antimicrobial effects of various endodontic irrigants on selected microorganisms. Int Endod J. 1999 Mar;32(2):99-102. doi: 10.1046/j.1365-2591.1999.00196.x. PMID 10371903
- [Result] Baumgartner JC, Cuenin PR. Efficacy of several concentrations of sodium hypochlorite for root canal irrigation. J Endod. 1992 Dec;18(12):605-12. doi: 10.1016/S0099-2399(06)81331-2. PMID 1298800
- [Result] Bystrom A, Sundqvist G. The antibacterial action of sodium hypochlorite and EDTA in 60 cases of endodontic therapy. Int Endod J. 1985 Jan;18(1):35-40. doi: 10.1111/j.1365-2591.1985.tb00416.x. No abstract available. PMID 3922900
- [Result] Fabricius L, Dahlen G, Sundqvist G, Happonen RP, Moller AJ. Influence of residual bacteria on periapical tissue healing after chemomechanical treatment and root filling of experimentally infected monkey teeth. Eur J Oral Sci. 2006 Aug;114(4):278-85. doi: 10.1111/j.1600-0722.2006.00380.x. PMID 16911098
- [Result] Hand RE, Smith ML, Harrison JW. Analysis of the effect of dilution on the necrotic tissue dissolution property of sodium hypochlorite. J Endod. 1978 Feb;4(2):60-4. doi: 10.1016/S0099-2399(78)80255-6. No abstract available. PMID 277629
- [Result] Harrison JW, Hand RE. The effect of dilution and organic matter on the anti-bacterial property of 5.25% sodium hypochlorite. J Endod. 1981 Mar;7(3):128-32. doi: 10.1016/S0099-2399(81)80127-6. No abstract available. PMID 6783724
- [Result] KAKEHASHI S, STANLEY HR, FITZGERALD RJ. THE EFFECTS OF SURGICAL EXPOSURES OF DENTAL PULPS IN GERM-FREE AND CONVENTIONAL LABORATORY RATS. Oral Surg Oral Med Oral Pathol. 1965 Sep;20:340-9. doi: 10.1016/0030-4220(65)90166-0. No abstract available. PMID 14342926
- [Result] Molander A, Warfvinge J, Reit C, Kvist T. Clinical and radiographic evaluation of one- and two-visit endodontic treatment of asymptomatic necrotic teeth with apical periodontitis: a randomized clinical trial. J Endod. 2007 Oct;33(10):1145-8. doi: 10.1016/j.joen.2007.07.005. PMID 17889679
- [Result] Moller AJ, Fabricius L, Dahlen G, Ohman AE, Heyden G. Influence on periapical tissues of indigenous oral bacteria and necrotic pulp tissue in monkeys. Scand J Dent Res. 1981 Dec;89(6):475-84. doi: 10.1111/j.1600-0722.1981.tb01711.x. PMID 6951246
- [Result] Peters LB, Wesselink PR. Periapical healing of endodontically treated teeth in one and two visits obturated in the presence or absence of detectable microorganisms. Int Endod J. 2002 Aug;35(8):660-7. doi: 10.1046/j.1365-2591.2002.00541.x. PMID 12196219
- [Result] Siqueira JF Jr, Rocas IN, Favieri A, Lima KC. Chemomechanical reduction of the bacterial population in the root canal after instrumentation and irrigation with 1%, 2.5%, and 5.25% sodium hypochlorite. J Endod. 2000 Jun;26(6):331-4. doi: 10.1097/00004770-200006000-00006. PMID 11199749
- [Result] Sjogren U, Figdor D, Persson S, Sundqvist G. Influence of infection at the time of root filling on the outcome of endodontic treatment of teeth with apical periodontitis. Int Endod J. 1997 Sep;30(5):297-306. doi: 10.1046/j.1365-2591.1997.00092.x. PMID 9477818
- [Result] Spangberg L, Engstrom B, Langeland K. Biologic effects of dental materials. 3. Toxicity and antimicrobial effect of endodontic antiseptics in vitro. Oral Surg Oral Med Oral Pathol. 1973 Dec;36(6):856-71. doi: 10.1016/0030-4220(73)90338-1. No abstract available. PMID 4208832
- [Result] Yesilsoy C, Whitaker E, Cleveland D, Phillips E, Trope M. Antimicrobial and toxic effects of established and potential root canal irrigants. J Endod. 1995 Oct;21(10):513-5. doi: 10.1016/s0099-2399(06)80524-8. PMID 8596073